CLINICAL TRIAL: NCT01667640
Title: Sector Irradiation Versus Whole Brain Irradiation After Resection of Singular or Solitary Brain Metastasis - a Prospective Randomized Monocentric Trial
Brief Title: Sector Irradiation Versus Whole Brain Irradiation for Brain Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Marcel Seiz-Rosenhagen MD, PD (Unknown); Meinhard Nevinny-Stickel MD, Prof. (Unknown); Christian F Freyschlag MD (Unknown); Günther Stockhammer MD, Prof. (Unknown); Bernhard Holzner MD, Doz (Unknown); Johannes Giesinger Mag (Unknown); Margarete Delazer MD, Prof. (Unknown); Thomas Bodner MD, MSc (Unknown); Claudius Thomé MD, Prof. (Unknown)
Responsible Party: Principal Investigator, Kerschbaumer Johannes, MD, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sektorradv_4.0_04-2012
Record Dates: First submitted 2012-08-07; First posted 2012-08-17 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Malignant Neoplasm to the Adult Brain
Keywords: Brain metastases; radiation; sector; singular; solitary; neurocognition
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- whole brain irradiation (Active Comparator): whole brain irradiation with 40 Gy, with fixation mask, radiation of the entire brain, skull base and meninges
  Interventions: Radiation: whole brain irradiation
- sector irradiation (Experimental): irradiation of the resection margin plus 5 mm safety margin with 30 Gy in 5 fractions
  Interventions: Radiation: sector irradiation

INTERVENTIONS:
Radiation: sector irradiation — Gross Tumor Volume (GTV) is defined as the visible margin of the resection on post- operative MRI and planning- CT-scan. The Clinical Treatment Volume (CTV) is the same as the GTV plus a 5 mm margin The Planning Treatment Volume (PTV) includes the CTV plus a 1mm margin.
  A non-invasive immobilization is used for the planning CT and treatment delivery with an accuracy of ≤ 1mm.
  Treatment planning will conform to ICRU 50/62 rules for coverage of GTV, CTV and PTV. Additionally, organs at risk are delineated according to the ICRU 62 rules.
  Treatment with radiotherapy will start 2 to 3 weeks after surgery. The prescribed dose for the PTV is 30 Gy in 5 fractions.
  Isodose distributions will be calculated through the target in three planes. Dose volume histograms will be reported.
  Arms: sector irradiation
Radiation: whole brain irradiation — For whole brain radiation the entire brain, the base of the skull and the meninges are included.
  Radiation is performed fractionated with 40 Gy. The caudal boundary of the radiation-target volume is between the 2. and the 3. cervical vertebra. The radiation is performed via two lateral, opposing and isocentric contra fields. The face/ventral skull is shielded with individual blocs or MLC.
  The used energy for the radiation fields should be between 6 and 16 MV. The specification point of the dose or the standardization point has to be chosen in that way that the point is in the middle of the target volume. The target volume is radiated within the tolerance range of 95% - 107 %. The maximum/minimum doses in the target volume and possible doses peaks are documented.
  Arms: whole brain irradiation

SUMMARY:
Microneurosurgical resection of intracerebral metastases leads to prolonged survival and relief of symptoms in selected patients.

To minimize the risk of intracranial recurrence whole brain irradiation has been established as standard adjuvant treatment in those patients. Sector irradiation resembles a brain - tissue - sparing method by focusing the irradiation in the area of the tumor bed and a surrounding 1mm security margin.

The aim of this study is to investigate whether adjuvant "sector""-irradiation following microsurgical resection is equal to adjuvant whole brain irradiation in terms of local control and superior to in terms of quality of life and neurocognitive deficits in a prospective randomized trial.

DETAILED DESCRIPTION:
Microneurosurgical resection of intracerebral metastases leads to prolonged survival and relief of symptoms in selected patients. Traditionally whole-brain irradiation is the treatment of choice following surgical resection. Whole brain irradiation has been the standard approach to minimize the risk of intracranial recurrence following resection of brain metastases. Almost 2 decades ago, Patchell et al. established the superiority of resection of solitary metastases followed by whole brain irradiation compared with whole brain irradiation alone with regard to survival, local control, and length of functional independence. A following study by the same group failed to show a survival advantage for the addition of whole brain irradiation compared to surgical resection alone in patients with a solitary intracranial metastasis, although the likelihood of local and distant recurrence and death from neurological causes were significantly reduced by whole brain irradiation. Due to potential delayed neurocognitive effects associated with whole brain irradiation, investigators have evaluated the use of partial brain irradiation in the form of stereotactic radiosurgery instead of whole brain irradiation after resection of brain metastases. They showed that despite whole brain irradiation means superior control of brain recurrence in sites other than the resection bed, stereotactic radiosurgery after resection resulted in equivalent survival times and neurological preservation. In a retrospective series of 52 patients Karlovits et al. could show that stereotactic radiosurgery following surgical resection leads to equal local control compared to standard whole brain irradiation.

Study objective

The aim of this study is to investigate whether adjuvant "sector" -irradiation following microsurgical resection is equal to adjuvant whole brain irradiation in terms of local control and superior to in terms of quality of life and neurocognitive deficits in a prospective randomized trial.

Hypothesis

1. Sector irradiation is equal to whole-brain irradiation in local tumor control after 3, 6, 12 and 36 months and
2. Sector irradiation" is superior to whole-brain irradiation in terms of quality of life and neurocognitive function

Patients and Methods

Patients with a single brain metastasis amenable to surgical resection fulfilling the inclusion criteria will be consecutively enrolled in this study. After microsurgical complete resection documented by early postoperative MRI within 72 hours and histological proven brain metastasis patients will be randomized in arm A or B. Radiotherapy will start after 14th postoperative day within 3 weeks postoperatively. Study arm A means postoperative sector irradiation (30Gy), study arm B includes standard whole brain radiotherapy (40Gy). Follow up MRI will be every 3 months. Neurocognitive evaluation will be performed before radiotherapy and 6 and 12 months postoperatively. In case of local recurrence or developing further metastases a cross over to whole brain radiotherapy or focal irradiation is possible.

ELIGIBILITY:
Inclusion Criteria:

* Solitary/singular brain metastasis
* Karnofsky Performance Index > 60%
* Stable extracranial disease /CUP
* Informed consent

Exclusion Criteria:

* Small cell lung cancer
* Squamous cell lung cancer
* HER2-negative breast cancer
* Deep-seated location (e.g. basal ganglia)
* Expected surgery related neurological deficit
* Tumor diameter < 3cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
local tumor control | time from date of randomization until the date of first documented progression, assessed up to 36 months

SECONDARY OUTCOMES:
distant brain metastasis | Time from date of randomization until the date of first documented progression elsewhere than the resection cavity, assessed at 3, 6, 12 and 36 months
time to clinical deterioration | Time from randomization to clinical deterioration, assessed by neurosurgeon in regular follow up visits at 3, 6, 12 and 36 months
local progression free survival | Time from randomization to the first documented tumor progressions in the resection cavity borders, assessed up to 36 months
quality of life | 3, 6, 12 and 36 months
  standardized assessment via "EORTC QLQ-C30/BN20" and the "FACT-Br" - questionary at 3, 6, 12 and 36 months after date of randomization
neurocognitive functions | 3, 6, 12 and 36 months postoperative
  Neurocognitive testing by independent neuropsychologist at 3, 6, 12 and 36 months after date of randomization
steroid dosage | 3, 6, 12 and 36 months postoperative
  Need of adjuvant steroid, assessed at 3, 6, 12 and 36 months after date of randomization
overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Seiz-Rosenhagen, MD, PD, Principal Investigator — Department of Neurosurgery, Medical University Innsbruck
Locations (1):
- Department of neurosurgery - Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Kerschbaumer J, Pinggera D, Holzner B, Delazer M, Bodner T, Karner E, Dostal L, Kvitsaridze I, Minasch D, Thome C, Seiz-Rosenhagen M, Nevinny-Stickel M, Freyschlag CF. Sector Irradiation vs. Whole Brain Irradiation After Resection of Singular Brain Metastasis-A Prospective Randomized Monocentric Trial. Front Oncol. 2020 Nov 24;10:591884. doi: 10.3389/fonc.2020.591884. eCollection 2020. PMID 33330076
- See also: Study center hompage. — http://neurochirurgie.uklibk.ac.at